CLINICAL TRIAL: NCT07289802
Title: Safety and Efficacy of the 3DMax MID Anatomical Mesh (BD, USA) in Laparoendoscopic Inguinal Hernia Repair: A Multicenter Prospective Observational Cohort Study
Brief Title: Safety and Efficacy of the 3DMax™ MID Anatomical Mesh (BD, USA) in Laparoscopic-endoscopic Inguinal Hernia Repair - Multicenter, Prospective Observational Study
Acronym: 3DMS
Status: Not yet recruiting | Type: Observational
Sponsor: Swissmed Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 3DMID-PL
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hernia, Inguinal
Keywords: Hernia; Mesh; Inguinal Hernia; Recurrence
MeSH Terms: conditions — Hernia, Inguinal; Hernia; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3DMax MID TAPP/TEP: Adult patients undergoing elective laparoendoscopic inguinal hernia repair (TAPP or TEP) with implantation of the 3DMax MID Anatomical Mesh (BD, USA) as part of routine clinical practice. No randomization or control group is used; all enrolled participants receive the same type of mesh according to the treating surgeon's standard technique.
  Interventions: Device: 3DMax MID Anatomical Mesh

INTERVENTIONS:
Device: 3DMax MID Anatomical Mesh — Implantation of a pre-shaped, medium-weight, macroporous polypropylene anatomical mesh (3DMax MID Anatomical Mesh, BD, USA) during elective laparoendoscopic inguinal hernia repair (TAPP or TEP) as part of routine clinical practice. No additional experimental procedures beyond standard surgical care are planned.
  Other Names: 3DMax MID

SUMMARY:
This is a multicenter, prospective, observational cohort study evaluating the safety and efficacy of the 3DMax MID Anatomical Mesh (BD, USA) in laparoendoscopic inguinal hernia repair. Adult patients undergoing elective transabdominal preperitoneal (TAPP) or totally extraperitoneal (TEP) repair will be enrolled and followed according to routine clinical practice.

The primary objective is to assess the inguinal hernia recurrence rate within 12 months after surgery. Secondary objectives include evaluation of postoperative pain, groin discomfort and foreign body sensation, as well as early and late postoperative complications.

All participating patients will receive the 3DMax MID Anatomical Mesh as part of standard care. No additional experimental procedures are planned. Clinical data will be collected at baseline and during predefined follow-up contacts (early postoperative period, 1 month, 3 months and 12 months) using standardized forms and patient interviews.

DETAILED DESCRIPTION:
Laparoendoscopic techniques such as transabdominal preperitoneal (TAPP) and totally extraperitoneal (TEP) repair are widely used for the treatment of inguinal hernia and are associated with faster recovery and lower rates of chronic pain compared with open repair in appropriately selected patients. Mesh reinforcement is a key component of these procedures. Three-dimensional, anatomically contoured meshes have been developed to improve conformability to the myopectineal orifice and to provide stable coverage of the inguinal region, potentially reducing the need for additional fixation and lowering the risk of chronic postoperative pain.

The 3DMax MID Anatomical Mesh (BD, USA) is a medium-weight, macroporous, pre-shaped polypropylene mesh designed specifically for inguinal hernia repair. Its three-dimensional configuration and recoil properties are intended to facilitate correct positioning and stable coverage of the inguinal anatomy during laparoendoscopic procedures.

This multicenter, prospective, observational cohort study will include consecutive adult patients undergoing elective TAPP or TEP inguinal hernia repair in participating centers, in whom the operating surgeon has decided to use the 3DMax MID Anatomical Mesh as part of routine practice. No randomization or control group is planned, and no interventions outside standard care will be performed.

Data will be collected from medical records and structured follow-up contacts (early postoperative check, approximately 30 days, 3 months and 12 months after surgery). The primary endpoint is hernia recurrence within 12 months. Secondary endpoints include postoperative pain, groin discomfort, foreign body sensation and early or late postoperative complications. Study data will be recorded in a standardized database and analyzed descriptively to characterize the safety profile and clinical performance of the 3DMax MID Anatomical Mesh in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Primary unilateral or bilateral inguinal hernia
* Scheduled for elective laparoendoscopic inguinal hernia repair (TAPP or TEP)
* Considered suitable for general anesthesia and laparoendoscopic approach by the treating surgeon
* 3DMax MID Anatomical Mesh planned for use as part of routine clinical care
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Age below 18 years
* Emergency surgery (e.g. incarcerated or strangulated hernia requiring urgent intervention)
* Contaminated or potentially contaminated surgical field
* Recurrent inguinal hernia in the same groin (previous repair with mesh or suture)
* Concomitant procedures or clinical situations in which the surgeon decides that a different mesh concept or technique is required
* Inability or unwillingness to comply with follow-up schedule (e.g. lack of telephone contact, severe cognitive impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with primary unilateral or bilateral inguinal hernia undergoing elective laparoendoscopic (TAPP or TEP) repair with implantation of the 3DMax MID Anatomical Mesh in participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Inguinal hernia recurrence rate at 12 months | 12 months after index surgery
  Proportion of patients with clinically and/or imaging-confirmed inguinal hernia recurrence within 12 months after the index laparoendoscopic repair with 3DMax MID Anatomical Mesh.

SECONDARY OUTCOMES:
Postoperative pain intensity (VAS 0-10) | 7-10 days, 30 days, 3 months and 12 months after surgery
  Postoperative pain intensity assessed using a 0-10 Visual Analog Scale (VAS) during early and late follow-up. Chronic pain will be defined as VAS ≥4 persisting beyond 3 months after surgery.
Early postoperative complications (≤30 days) | Up to 30 days after surgery
  Incidence of early postoperative complications within 30 days after surgery, including wound infection, hematoma, seroma, urinary retention, bleeding, and other mesh- or procedure-related adverse events.
Late postoperative complications (>30 days to 12 months) | From >30 days to 12 months after surgery
  Incidence of late postoperative complications occurring between 30 days and 6 months after surgery, including chronic groin pain, mesh-related complications, and reoperations in the operated groin.
Groin discomfort and foreign body sensation | 7-10 days, 30 days, 3 months and 12 months after surgery
  Patient-reported groin discomfort, stiffness and foreign body sensation in the operated region, assessed using standardized questions or Likert-type scales during follow-up contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Śmietański, Prof., Study Chair — LUX MED Hospital in Gdańsk; Mateusz Zamkowski, MD, PhD, Principal Investigator — LUX MED Hospital in Gdańsk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zamkowski M, S Mietanski M, Franczak P, Gorski D, Grabias J, Janik M, Krol A, Mitura K, Medras O, Nawacki L, Romanczuk M, Rymkiewicz P, Saluk S, Sroczynski P, Sulkowski L, Wieczorek D, Wlodarczyk M. MEsh FIxation STudy in Laparoendoscopic Repair of M3 Inguinal Hernias: Multicenter, Double-blind, Randomized Controlled Trial-MEFISTO Trial. Ann Surg. 2025 Jun 1;281(6):921-927. doi: 10.1097/SLA.0000000000006669. Epub 2025 Feb 13. PMID 39945075
- [Background] Zamkowski M, Tomaszewska A, Lubowiecka I, Karbowski K, Smietanski M. Is mesh fixation necessary in laparoendoscopic techniques for M3 inguinal defects? An experimental study. Surg Endosc. 2023 Mar;37(3):1781-1788. doi: 10.1007/s00464-022-09699-5. Epub 2022 Oct 13. PMID 36229552
- [Background] Zamkowski M, Smietanski M. MEsh FIxation in Laparoendsocopic Repair of Large M3 inguinal hernias: multicenter, double-blinded, randomized controlled trial-study protocol for a MEFI Trial. Trials. 2023 Sep 5;24(1):572. doi: 10.1186/s13063-023-07601-9. PMID 37670376
- [Background] Mateusz Zamkowski, Agnieszka Tomaszewska, Izabela Lubowiecka, Krzysztof Karbowski, Michał Putko, Maciej Śmietański. Mechanical stability of new-generation meshes for M3 inguinal hernia repair: experimental pressure chamber testing of SWING-Mesh® and 3DMax™ MID Anatomical Mesh DOI: 10.20452/wiitm.2025.17990 Published online: October 29, 2025